CLINICAL TRIAL: NCT01713998
Title: Evaluation of the Ulthera® System for Lifting and Tightening the Face and Neck With Lower Energy Settings
Brief Title: Treatment of the Face and Neck With Lower Ulthera System Energy Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-300
Record Dates: First submitted 2012-10-15; First posted 2012-10-25 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Subjects will receive an increased density Ulthera System Treatment over the full face but with the energy turned down to the second highest level of four possible energy settings on one side of the face.
  Interventions: Device: Ulthera System Treatment
- Group B (Active Comparator): Subjects will receive an increased density guideline Ulthera System Treatment over the full face but with the energy turned down to the lowest level of four possible energy settings on one side of the face.
  Interventions: Device: Ulthera System Treatment
- Group C (Active Comparator): Subjects will receive an increased density guideline Ulthera System Treatment over the full face with the exception that a 4 MHz transducer will be used on the upper face in place of a7 MHz transducer, with the energy turned down to the lowest level of four possible energy settings.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 60 subjects will be enrolled. Enrolled subjects will receive one Ulthera® treatment on the face and neck. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This trial is a prospective, single-site, double-blinded, randomized, split-face design. Subjects will be randomized to one of three treatment groups, receiving treatment using different energy levels. Global Aesthetic Improvement Scale scores and patient satisfaction questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years.
* Subject in good health.
* Skin laxity on the face and neck

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the face or neck.
* Excessive skin laxity on the face or neck.
* Significant scarring in areas to be treated.
* Open wounds or lesions in the area to be treated.
* Severe or cystic acne on the area to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Gitt, MD, Principal Investigator — Ulthera, Inc
Locations (1):
- Ulthera, Inc., Mesa, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-seven subjects were enrolled, randomized, and treated. The first subject treated on 10/4/2011; the last subject treated on 2/13/12; the last follow-up was 10/11/12.
  Enrolled subjects were randomized to one of three study groups (Group A, B, or C).
Groups:
- Group A: Subjects received an increased density guideline treatment over the full face but with the energy reduced to the second highest level of four possible energy settings on one side of the face.
- Group B: Subjects received an increased density guideline treatment over the full face but with the energy reduced to the lowest level of four possible energy settings on one side of the face.
- Group C: Subjects received an increased density guideline treatment over the full face. The upper face treatment was provided in a split-face treatment using the 4 MHz transducer at no higher than the second highest energy setting on one side of the upper face and the 7 MHz transducer at the highest energy setting on other side of the upper face.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 16 | 15 | 16
Completed | 13 | 15 | 14
Not Completed | 3 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Subjects received Ultherapy® treatment using standard (highest) energy settings on one side of the face, and energy adjusted down to the second highest level of four possible energy settings on the contralateral side of the face.
- Group B: Subjects received Ultherapy® treatment using standard (highest) energy settings on one side of the face, and energy adjusted down to the lowest level of four possible energy settings on the contralateral side of the face.
- Group C: Subjects received Ultherapy® treatment using standard (highest) energy settings on both sides of the lower face and neck. On the upper face (brow), the 4-4.5mm transducer used at the second highest energy setting on one side of the upper face and the 7-4.5mm transducer at the standard (highest) energy setting on the contralateral side of the upper face.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 16 | 15 | 16 | 47
Age, Continuous [Mean (Full Range); unit: years] | 54 [37 to 64] | 55 [42 to 64] | 51 [36 to 64] | 53 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 14 | 45
  Male | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 15 | 14 | 14 | 43
  Hispanic/Latino | 0 | 1 | 1 | 2
  Asian | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 16 | 47
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 24 [20 to 29] | 24 [19 to 28] | 24 [20 to 29] | 24 [19 to 29]
Fitzpatrick Skin Type [Number; unit: participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  participants
    Skin Type I | 0 | 1 | 0 | 1
    Skin Type II | 10 | 5 | 5 | 20
    Skin Type III | 6 | 7 | 10 | 23
    Skin Type IV | 0 | 2 | 1 | 3
    Skin Type V | 0 | 0 | 0 | 0
    Skin Type VI | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjects' Assessment of Pain During Treatment With Lower Energy Settings
Description: Subjects' sensory response to the Ulthera treatment exposures were recorded using a validated Numeric Rating Scale (NRS,0-10), for each anatomical region treated and energy settings used, with 0 representing no pain and 10 representing the worst pain possible.
  Pain scores were collected in a consistent manner, following treatment of each section of the face and neck on both sides (submental, submandibular, cheek, periorbital, infraorbital, and forehead), and for each transducer used. Split-face comparisons of pain scores obtained during study treatment by research staff blinded to the energy settings used were completed.
Time Frame: Participants were assessed for the duration of study treatment, an average of 75 minutes
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Group C: Subjects received a standard Ultherapy® treatment using the (standard) highest energy settings on both sides of the lower face and neck. On the upper face (brow), the 4 MHz transducer was used at the (adjusted)second highest energy setting on one side of the upper face, and the 7 MHz transducer at the (standard) highest energy setting on the contralateral side of the upper face. For this outcome measure, only pain score data reported for the brow regions (using standard versus adjusted energy settings) were included.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 16 | 15 | 16
units on a scale
  Standard Energy | 4.5 [1 to 10] | 6.0 [1 to 10] | 5.6 [3 to 10]
  Adjusted Energy | 3.7 [1 to 9] | 3.7 [0 to 8] | 5.9 [3 to 10]

2. Primary Outcome: Overall Improvement in Skin Laxity on the Face and Neck
Description: A split-face comparison of improvement in overall lifting and tightening of skin was completed by three masked assessors. Pre-treatment and 90 days post-treatment photos from 45 subjects who returned for their 90-day follow-up visit were reviewed, assessing for improvement in skin laxity, i.e., lifted and tightened skin in the areas treated using treatment energy settings based on subjects' assigned study group.
Time Frame: 90 days post-treatment
Measure: Number; unit: Participants
Groups:
- Group C: Subjects received a standard Ultherapy® treatment using the (standard) highest energy settings on both sides of the lower face and neck. On the upper face (brow), the 4 MHz transducer was used at the (adjusted) second highest energy setting on one side of the upper face, and the 7 MHz transducer at the (standard) highest energy setting on the contralateral side of the upper face. For Group C, the standard energy side is defined as the upper face side treated with the 7 MHz transducer at the highest energy setting and the corresponding lower face side; the adjusted energy side is defined as the upper face side treated with 4 MHz transducer at the second highest energy setting and the corresponding lower face side.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
Participants | 6 | 6 | 6

3. Secondary Outcome: Quantitative Assessment of Brow Lift at 90 Days Post-treatment
Description: Quantitative assessment and analysis of brow lift from baseline to 90 days post-treatment was completed comparing brow lift achieved using standard energy settings compared to adjusted energy settings. The number of subjects with 1 mm or more brow lift is reported. Note: Because the submental region was treated using standard energy settings in all study groups, a quantitative analysis of lift in this region between the study groups would most likely not be informative, and therefore was not completed.
Time Frame: 90 days post-treatment
Measure: Number; unit: Participants
Groups:
- Group C: Subjects received a standard Ultherapy® treatment using the (standard) highest energy settings on both sides of the lower face and neck. On the upper face (brow), the 4-4.5mm transducer was used at the (adjusted)second highest energy setting on one side of the upper face, and the 7-4.5mm transducer at the (standard) highest energy setting on the contralateral side of the upper face. For Group C, the standard energy side is defined as the upper face side treated with the 7-4.5mm transducer at the highest energy setting and the corresponding lower face side; the adjusted energy side is defined as the upper face side treated with 4-4.5mm transducer at the second highest energy setting and the corresponding lower face side.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Standard Energy | 2 | 5 | 2
  Adjusted Energy | 2 | 3 | 6

4. Secondary Outcome: Subject Assessment of Improvement at 90 Days Post-treatment
Description: Subjects completed a Patient Assessment Questionnaire at 90 days post-treatment by referring to their image in a mirror, their 90-day post-treatment photos, and their pre-treatment photos, and reporting if any improvement was noted on the right and left sides of their face and neck.
Time Frame: 90 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 15 | 15
percentage of participants
  Standard Energy | 86 | 80 | 93
  Adjusted Energy | 93 | 80 | 87

5. Secondary Outcome: Subject Assessment of Improvement at 180 Days Post-treatment
Description: Subjects completed a Patient Assessment Questionnaire at 180 days post-treatment by referring to their image in a mirror, their 180-day post-treatment photos, and their pre-treatment photos, and reporting if any improvement was noted on the right and left sides of their face and neck.
Time Frame: 180 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 15 | 14
percentage of participants
  Standard Energy | 77 | 73 | 86
  Adjusted Energy | 75 | 80 | 79

ADVERSE EVENTS:
Groups:
- Study Population: Includes all subjects meeting entrance criteria, consented for participation, enrolled and randomized.
Arm/Group | Study Population
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No